CLINICAL TRIAL: NCT06928259
Title: Clinical Relevance of Drug-drug Interactions (DDI) With the Currently Used Direct-acting Antiviral Therapy (DAA) Against Hepatitis C Virus (HCV)
Brief Title: Drug-Drug Intercations and Direct Acting Antiviral Agents Against HCV
Status: Recruiting | Type: Observational
Sponsor: University of Seville (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Juan Macías, Profesor de Medicina, University of Seville
Other Study IDs: CO-ES-342-7138
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: HCV Infection
Keywords: HCV; SOF/VEL; GLE/PIB; drug-drug interactions
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SOF/VEL: Treatment with SOF/VEL (n=485)
- GLE/PIB: Treatment with GLE/PIB (n=243)

SUMMARY:
Background: Currently used direct-acting antivirals (DAA) share pharmacokinetic pathways with many comedications commonly used in patients with chronic hepatitis C virus (HCV) infection, therefore drug-drug interactions (DDI) might exist. Although extensive (DDI) verification is recommended by most clinical practice guidelines, real-world studies have shown that approximately one-tenth of patients on DAA therapy also take concomitant medication with the potential for significant interactions. Despite the risk of significant DDI when patients are administered DAA and a concomitant medication, to date, there is very little information on whether these interactions translate into changes in the toxicity or efficacy of any involved DAA or comedication in clinical practice. Clarifying this issue is a critical point, as the DDI profile of the currently used DAA is not the same, with SOF/VEL showing a lower risk of significant DDI than GLE/PIB. Thus the objective of this study is to compare the percentage of comedication switch, withdrawal, or dose reduction at treatment initiation and during treatment with GLE/PIB or SOF/VEL.

Methods: The patients will be enrolled from the GEHEP 001/HEPAVIR cohort. "The HEPAVIR-DAA cohort (NCT02057003)", includes HIV/HCV-coinfected patients, and "the GEHEP-MONO cohort (NCT02333292)", that includes HCV mono-infected individuals, are ongoing prospective multicenter cohorts of patients receiving DAA combinations prescribed in clinical practice, outside clinical trials. Main Study End Point will be the frequency of comedication switch, withdrawal or dose reduction at treatment initiation (index date) and during treatment with GLE/PIB or SOF/VEL.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naive patients who received therapy with GLE/PIB or SOF/VEL between April 1st, 2018, and July 1st, 2023, receiving ≥ 1 comedication or recreational drug.
2. Attended in a hospital with electronic clinical records allowing access to all clinical visits and prescribed medications, both in all hospitals and in primary care institutions of the corresponding Spanish region during the study period.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. HCV treatment-experienced patients will be excluded.
2. Patients without any comedication or recreational drug use
3. Those who have attended private health care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients will be enrolled from the GEHEP 001/HEPAVIR cohort. "The HEPAVIR-DAA cohort (NCT02057003)", includes HIV/HCV-coinfected patients, and "the GEHEP-MONO cohort (NCT02333292)", that includes HCV mono-infected individuals, are ongoing prospective multicenter cohorts of patients receiving DAA combinations prescribed in clinical practice, outside clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Main Study End Point | 90 days before treatment, 8-12 weeks of treatment, 24 weeks post treatment
  Frequency of comedication switch, withdrawal or dose reduction at treatment initiation (index date) and during treatment with GLE/PIB or SOF/VEL.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Unidad de Enfermedades Infecciosas Hospital Universitario Puerto Real., Cadiz
  - Unidad de Enfermedades Infecciosas. Hospital Universitario Reina Sofía de Córdoba., Córdoba
  - Unidad de Enfermedades Infecciosas. Hospital Universitario Juan Ramón Jiménez., Huelva
  - Departamento de Medicina. Universidad de Sevilla Hospital Universitario Virgen de Valme., Seville

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR